CLINICAL TRIAL: NCT04562870
Title: A Phase 2, Randomized, Open-Label, Multicenter Study to Evaluate Safety and Efficacy of Single Agent Selinexor Versus Treatment of Physician's Choice in Patients With Previously Treated Myelofibrosis
Brief Title: A Study to Evaluate Single Agent Selinexor Versus Physician's Choice in Participants With Previously Treated Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-MF-035; 2020-003809-60 (EudraCT Number); 2024-513605-31-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-09; First posted 2020-09-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Selinexor; Total Symptom Score; Spleen Volume Reduction; Anemia response; TSS50; SVR35; SVR25; KPT-330; JAK1; JAK2; XPOVIO; SINE; XPORT-MF-035; Karyopharm
MeSH Terms: conditions — Primary Myelofibrosis | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm S: Selinexor (Experimental): Participants with MF who had previously received at least 6 months of treatment with JAK 1/2 inhibitor will receive a dose of selinexor 80 mg for first 2 cycles followed by selinexor 60 mg once weekly (QW) in subsequent cycles orally on Days 1, 8, 15, and 22 of each 28-day cycle to participants on Arm S.
  Interventions: Drug: Selinexor
- Arm PC: Physician's Choice Treatment (Active Comparator): Participants with MF who had previously received at least 6 months of treatment with JAK 1/2 inhibitor will receive Physician's choice treatment which will be administered as per clinical practice.
  Interventions: Other: Physician's Choice Treatment

INTERVENTIONS:
Drug: Selinexor — Unit Dose Strength: 20 mg; Dose Formulation: Tablet; Dosage Level: 60 or 80 mg, QW; Route of Administration: Oral
  Arms: Arm S: Selinexor
Other: Physician's Choice Treatment — Physician's choice treatment may include ruxolitinib retreatment, fedratinib, chemotherapy (e.g., hydroxyurea), anagrelide, corticosteroid, hematopoietic growth factor, immunomodulatory agent, androgen, interferon (all as per clinical practice) and may include supportive care only with no MF treatment; no investigational therapies are allowed.
  Arms: Arm PC: Physician's Choice Treatment

SUMMARY:
This is a Phase 2, multicenter, two-arm, open-label study to evaluate the safety and efficacy of selinexor versus treatment per physician's choice (PC) in participants with myelofibrosis (MF) who had at least 6 months of treatment with a Janus kinase (JAK)1/2 inhibitor. Study participants will be randomized in a 1:1 ratio to either receive selinexor or physicians' choice of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary MF or post-essential thrombocythemia (ET) or post-polycythemia (PV) MF according to the 2016 World Health Organization (WHO) classification of myeloproliferative neoplasms (MPN), by the most recent local pathology report.
* Previous treatment with JAK inhibitors for at least 6 months.
* Measurable splenomegaly during the screening period as demonstrated by spleen volume of ≥450 centimeter cube (cm^3) by magnetic resonance imaging (MRI) or computerized tomography (CT) scan.
* Relapsed, Refractory or Intolerant to JAK inhibitors as defined as meeting one of the criteria below:

  * less than (<) 35% spleen volume reduction by MRI or CT-scan (from baseline) or
  * <50% decrease in spleen size by palpation (from baseline) or an increase of at least 3 cm with the spleen at least 5 cm below the left costal margin or
  * Spleen volume increase greater than (>) 25% from nadir or a return to within 10% of baseline after any initial response or
  * Treatment with JAK inhibitor was complicated by development of red blood cells (RBC) transfusion requirement (2 units per month for 2 month); or grade 3 thrombocytopenia, anemia, hematoma/hemorrhage; or grade 2 non-hematologic toxicity while on JAK inhibitors
* Participants ≥18 years of age.
* Eastern Cooperative Oncology Group (ECOG) less than or equal to (≤) 2.
* Platelet count ≥75*10^9 per liter (/L).
* Absolute neutrophil count (ANC) ≥1.5*10^9/L.
* Serum direct bilirubin ≤1.5*upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5*ULN.
* Calculated creatinine clearance (CrCl) >15 milliliter (mL)/minute (min) based on the Cockcroft and Gault formula.
* Participants with active hepatitis B virus (HBV) are eligible if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 International Units (IU)/mL.
* Participants with untreated hepatitis C virus (HCV) are eligible if there is a documentation of negative viral load per institutional standard.
* Participants with history of human immunodeficiency virus (HIV) are eligible if they have cluster of differentiation 4 (CD4)+ T-cell counts ≥350 cells/microliter (mcL), negative viral load per institutional standard, and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year.
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective methods of contraception throughout the study and for at least 90 days after the last dose of selinexor, or for the duration as stated on the label (SmPC/USPI) for those on the comparator drug (physician's choice arm). Childbearing potential excludes: Age >50 years and naturally amenorrhoeic for >1 year, or previous bilateral salpingo-oophorectomy, or hysterectomy.
* Male participants who are sexually active must use highly effective methods of contraception throughout the study and for at least 90 days after the last dose of selinexor, or for the duration as stated on the label (SmPC/USPI) for those on the comparator drug (physician's choice arm). Male participants must agree not to donate sperm during the study treatment period.
* Participants must sign written informed consent in accordance with federal, local and institutional guidelines.

Exclusion Criteria:

* >5% blasts in peripheral blood or >10% blasts in bone marrow (i.e., accelerated phase).
* Previous treatment with selinexor or other exportin 1 (XPO1) inhibitors.
* Use of any standard or experimental anti-MF therapy <21 days prior to Cycle 1 Day 1 (hydroxyurea or growth factors are allowed).
* Impairment of gastrointestinal (GI) function or GI disease that could significantly alter the absorption of selinexor (Example: vomiting, or diarrhea that is Common Terminology Criteria for Adverse Events (CTCAE) grade >1).
* Received strong cytochrome P450 3A (CYP3A) inhibitors ≤7 days prior to selinexor dosing or strong CYP3A inducers ≤14 days prior to selinexor dosing.
* Major surgery <28 days prior to cycle 1 day 1 (C1D1).
* Uncontrolled (ie, clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable (including parenteral).
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the participants safety, prevent the participant from giving informed consent, or being compliant with the study procedures.
* Female participants who are pregnant or lactating.
* Participants with contraindications to use of selinexor or all the drugs intended to be used in the comparative treatment arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Spleen Volume Reduction of Greater Than or Equal to (≥) 35 Percent (%) (SVR35) | From Baseline up to Week 24

SECONDARY OUTCOMES:
Percentage of Participants with Total Symptom Score Reduction of ≥50% (TSS50) Measured by Myelofibrosis Symptom Assessment Form (MFSAF) V4.0, Based on Local Assessment | From Baseline up to Week 24
Percentage of Participants with Spleen Volume Reduction of ≥25% (SVR25) | From Baseline up to Week 24
Overall Survival (OS) | From Baseline up to 12 months after end of treatment (approximately 48 months)]
Percentage of Participants with Anemia Response Assessed by International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) | From Baseline up to 28 days after last dose (approximately 48 months)
Duration of Spleen Volume Reduction of ≥35% (SVR35) | From Baseline up to Week 24
Duration of Spleen Volume Reduction of ≥25% (SVR25) | From Baseline up to Week 24
Duration of Total Symptom Score is ≥50% (TSS50) Based on Local Assessment | From Baseline up to Week 24
Overall Response Rate (ORR) Assessed by IWG-MRT | From Baseline up to 28 days after last dose (approximately 48 months)
Number of Participants With Treatment-emergent Adverse Events (TEAEs) by Severity Grade ≥3, Serious Adverse event (SAEs), and AEs Leading to Treatment Discontinuation | From first dose of study treatment up to 30 days after end of treatment (approximately 48 months)
Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration-time Curve (AUC) of Selinexor | Cycle 2 Day 1: 1, 2, 4, and 6 hours post-dose; Cycle 2 Day 2: at 24 hours post-dose (each cycle is 28 days)
PK Parameter: Maximum Plasma Concentration (Cmax) of Selinexor | Cycle 2 Day 1: 1, 2, 4, and 6 hours post-dose; Cycle 2 Day 2: at 24 hours post-dose (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (4):
  - The Oncology Institute of Hope and Innovation, Pasadena, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Illinois Cancer Specialist, Niles, Illinois
  - Texas Oncology - Northeast Texas, Tyler, Texas
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Suzhou University -The First Affiliated Hospital, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Sir Run Run Shaw Hospital - Zhejiang University School of Medicine, Hangzhou, Zhejiang
- France (2):
  - Institut de Cancéro-Hématologie, Brest, Brittany Region
  - Centre Hospitalier Universitaire d'Angers (CHU Angers), Angers
- University General Hospital "ATTIKON", Athens, Attica, Greece
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola, Forlì-Cesena
  - Università degli Studi di Firenze - Azienda Ospedaliero - Universitaria Careggi - Dipartimento di medicina sperimentale e clinica, Florence
  - Azienda Unita Sanitaria Locale Latina - Ospedale Santa Maria Goretti, Latina
  - University of Perugia Department of Medicine Hematology Section, Perugia
  - Asst Settelaghi, Ospedale Di Circolo E Fondazione Macchi, Varese
- Pratia Onkologia Katowice, Katowice, Poland
- Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided